CLINICAL TRIAL: NCT06058416
Title: The Immunogenicity and Safety of Different Vaccination Interval of Inactivated Hepatitis A Vaccine in People Aged 18-50 Years, a Phase IV Clinical Trial
Brief Title: Immunogenicity and Safety of Hepatitis A Among People Aged 18-50 Years Old
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Liaoning Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HAV-MA4001-LN
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis A
Keywords: immunogenicity and safety of vaccine; hepatitis A vaccine; vaccination schedule
MeSH Terms: conditions — Hepatitis A; Hepatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- immunogenicity group with vaccination interval of 6 month (Other)
  Interventions: Biological: Healive (hepatitis A vacine(human diploid cell), inactivated)
- immunogenicity group with vaccination interval of 18 month (Other)
  Interventions: Biological: Healive (hepatitis A vacine(human diploid cell), inactivated)
- immunogenicity group with vaccination interval of 36 month (Other)
  Interventions: Biological: Healive (hepatitis A vacine(human diploid cell), inactivated)
- immunogenicity group with vaccination interval of 60 month (Other)
  Interventions: Biological: Healive (hepatitis A vacine(human diploid cell), inactivated)
- safety observation group (Other)
  Interventions: Biological: Healive (hepatitis A vacine(human diploid cell), inactivated)

INTERVENTIONS:
Biological: Healive (hepatitis A vacine(human diploid cell), inactivated) — The hepatitis A vaccine contains 500 SU inactivated hepatitis A virus per dose in 1mL of aluminum hydroxide solution.
  For anti-HAV antibody-negative participants, two dose of hepatitis A vaccine will be given with vaccination interval of 6 month, 18 months, 36 months, and 60 months, respectively.

SUMMARY:
This study is conducted among people aged 18-50 in Dandong City, an area with a high incidence of hepatitis A in recent years. 1000 qualified pariticipants with signed informed consent will be screened for anti-HAV antibodies by collecting blood sample of 3ml. One dose of hepatitis A vaccine will be administrated to all the pariticipants. Negative anti-HAV antibodies-negative subjects will recieve the second dose of hepatitis A vaccination, and 400 of them will be randomly selected and assigned to 4 groups with different interval of vaccination(6 month, 18 months, 36 months and 60 months). Blood samples will be collected before vaccination of each dose and on 28 days after each dose of vaccination to anti-HAV antibody test. Safety data will be collected within 28 days after each vaccination with a smartphone mini-program.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50;
* Adults can understand and sign the informed consent form voluntarily;
* Adults can provide valid and legal identity certificate.

Exclusion Criteria:

* A history of hepatitis A infection;
* Previously vaccinated with inactivated hepatitis A vaccine, live attenuated hepatitis A vaccine, or hepatitis A and B combined vaccine;
* Allergic constitution or have severe allergic reaction to vaccines in the past (such as acute allergic reaction, angioedema, dyspnea, etc.);
* Pregnant women and lactating women;
* People suffering from uncontrolled epilepsy and other serious neurological diseases (such as transverse myelitis, Guillain-Barré syndrome, demyelinating diseases, etc.);
* Patients with fever during vaccination, or acute exacerbation of chronic diseases, or patients with uncontrolled severe chronic diseases, or suffering from acute diseases;
* Received other research drugs within 30 days before vaccination with the experimental vaccine;
* Have received a live attenuated vaccine within 14 days before vaccination with the experimental vaccine;
* Have received subunit or inactivated vaccine within 7 days before vaccination with experimental vaccine;
* Other conditions that are not suitable for vaccination judged by the researcher.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1092 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-03-17 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The seroconversion rate of anti-HAV antibody 28 days after two dose of vaccination of hepatitis A vaccine with an interval of 6 month | 28 days after two dose of vaccination of hepatitis A vaccine
Incidence of adverse reaction within 28 days after one dose of vaccination | 28 days after one dose of vaccination

SECONDARY OUTCOMES:
The seroconversion rate of anti-HAV antibody 28 days after two dose of vaccination of hepatitis A vaccine with an interval of 18 month, 36 months, and 60 months | 28 days after two dose of vaccination
The seropositive rate, GMC and GMI of anti-HAV antibody 28 days after two dose of vaccination of hepatitis A vaccine with an interval of 6 months, 18 month, 36 months, and 60 months | 28th day after two dose of vaccination
The seropositive rate, GMC and GMI of anti-HAV antibody 28 days after one dose of vaccination of hepatitis A vaccine with an interval of 6 months, 18 month, 36 months, and 60 months | 28 days after one dose of vaccination
The seropositive rate, GMC and GMI of anti-HAV antibody 28 days after two dose of vaccination of hepatitis A vaccine with an interval of 6 months, 18 month, 36 months, and 60 months among people with underlying conditions | 28 days after two dose of vaccination
The seropositive rate of anti-HAV antibody before vaccination | before vaccination
Incidence of adverse reaction within 7 days after one dose of vaccination | 7 days after one dose of vaccination
Incidence of adverse reaction within 28 days after two dose of vaccination | 28 days after two dose of vaccination
Incidence of adverse reaction within 28 days after one dose of vaccination among different group of people | 28 days after one dose of vaccination among

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Center for Disease Control and Prevention, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu XE, Chen HY, Liao Z, Zhou Y, Wen H, Peng S, Liu Y, Li R, Li J, Zhuang H. Comparison of Immunogenicity Between Inactivated and Live Attenuated Hepatitis A Vaccines Among Young Adults: A 3-Year Follow-up Study. J Infect Dis. 2015 Oct 15;212(8):1232-6. doi: 10.1093/infdis/jiv213. Epub 2015 May 12. PMID 25969561
- [Background] Iwarson S, Lindh M, Widerstrom L. Excellent booster response 4 to 8 years after a single primary dose of an inactivated hepatitis A vaccine. J Travel Med. 2004 Mar-Apr;11(2):120-1. doi: 10.2310/7060.2004.17079. No abstract available. PMID 15109480
- See also: ACIP — https://www.cdc.gov/mmwr/preview/mmwrhtml/rr5507a1.htm#tab2
- See also: WHO position paper on hepatitis A vaccines-October2022 — https://www.who.int/publications/i/item/who-wer9740-493-512